CLINICAL TRIAL: NCT03693651
Title: Prospective Study of the Quality of Sleep of Parents of Premature Children Hospitalized in Neonatology Compared to Parents of Full-term Children in Maternity
Brief Title: Study of the Quality of Sleep of Parents of Premature Children Compared to Parents of Full-term Children
Acronym: SLEEP-PP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: SLEEP-PP (29BRC18.0079)
Record Dates: First submitted 2018-08-23; First posted 2018-10-03 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-01

CONDITIONS: Prematurity; Parenting; Sleep Deprivation
MeSH Terms: conditions — Premature Birth; Sleep Deprivation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parent of a Premature infant / PP: self-report questionnaire that assesses sleep quality (The Pittsburgh Sleep Quality Index (PSQI)) filled at 1 month, 3 months and 6 months from child birth.
- Parent of a baby born on time / PT: self-report questionnaire that assesses sleep quality (The Pittsburgh Sleep Quality Index (PSQI)) filled at 1 month, 3 months and 6 months from child birth.

SUMMARY:
This study evaluate the incidence of sleep disorders in parents of premature children hospitalized in unit care of neonatalogy or intensive unit care of neonatalogy, compared to parents of full-term child in maternity.

ELIGIBILITY:
Inclusion Criteria:

* Couple of parents of children born before term (between 25 and 36 weeks) and hospitalized at the CHRU de Brest.
* Parents of healthy full-term children born at Brest CHRU (> 37 weeks) without neonatal hospitalization.
* Having formulated their agreement

Exclusion Criteria:

* Parents whose child died in the neonatal period.
* Couple whose one parents are minors at the birth of the child.
* Parents of children with malformation and /or genetic anomaly.
* Parents with known addiction, depressive syndrome or known psychiatric condition before birth.
* Single parent family.
* Non-French speaking parents.
* Refusal of participation of one of the parents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Couple of Parents of child born at the CHRU of Brest (full-term in maternity or premature child (25-36 weeks) hospitalized in maternity, neonatalogy or unity of intensive neonatal care).
  Both Parents will be included, each of them will have to fill the PSQI at 1, 3 and 6 months from the child birth.
Sampling Method: Non-Probability Sample
Enrollment: 306 (Estimated)
Dates: Start 2018-06-14 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Scale Pittsburgh Sleep Quality Index (PSQI) | 6 months from child Birth
  Online self-report questionnaire that assesses sleep quality filled at 1 month, 3 months and 6 months from child birth.
  This questionnaire has been validated to assess the presence of sleep disorders.
  It includes 19 questions that combine to evaluate 7 components of sleep, each evaluated from 0 to 3 (0 = no difficulty, 3 = severe difficulty).
  A total score greater than 5 indicates a sleep disorder.

SECONDARY OUTCOMES:
The Pittsburgh Sleep Quality Index (PSQI) | 1 month from child birth
  Online self-report questionnaire that assesses sleep quality filled at 1 month, 3 months and 6 months from child birth.
The Pittsburgh Sleep Quality Index (PSQI) | 3 months from child birth
  Online self-report questionnaire that assesses sleep quality filled at 1 month, 3 months and 6 months from child birth.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No